CLINICAL TRIAL: NCT03273777
Title: Comparison of Skin Incision Skewness With or Without Previous Measurement and Drawing of the Incision Line at Cesarean Section - a Randomized Controlled Trial
Brief Title: Skin Incision Skewness at Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Heinrich Husslein, Ass.-Prof., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1641_2016
Record Dates: First submitted 2017-06-06; First posted 2017-09-06 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Cesarean Section
Keywords: Cesarean section; Skin incision; Skewness; Line drawing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drawing of an incision line (Experimental): An incision line of 14 cm will be drawn using a conventional surgical ruler and pen before skin incision.
  Interventions: Procedure: Drawing of an incision line
- No drawing of an incision line (No Intervention): Skin incision will be carried out without previous drawing of an incision line.

INTERVENTIONS:
Procedure: Drawing of an incision line — Drawing of an incision line prior to skin incision at cesarean section
  Arms: Drawing of an incision line

SUMMARY:
Skin incision skewness, incision length on both sides of the midline and patient's perception of the scar after cesarean section will be compared between the following two groups: (1) Drawing of an incision line prior to skin incision and (2) no drawing of an incision line.

DETAILED DESCRIPTION:
Some aspects of the surgical techniques employed during cesarean section have already been evaluated in regards to possible improvements of cosmetic outcome, such as the use of different skin closure materials or whether subcutaneous fat suture closure leads to better results than non-closure. Another point to be considered is the skewness of the scar. Many surgeons make the skin incision based on their experience without prior measurement and drawing of an incision line. However, following a predefined incision line may reduce the rate of skew incisions. Therefore, this study aims to compare these two approaches to the skin incision.

Participating women will be recruited at the Department of Obstetrics and Gynecology of the Medical University of Vienna. They will be included into the study after written informed consent and will be randomized into one of the two groups (drawing of an incision line prior to skin incision versus no drawing of an incision line) on the day of cesarean section.

Skewness of the skin incision in each group will be assessed after cesarean section. Furthermore, it will be determined whether there are any differences in the incision length on both sides of an imaginary line from the umbilicus to the clitoris between these two techniques. Additionally, patient's perception of the scar before discharge from hospital will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* First cesarean section

Exclusion Criteria:

* Performance of an acute cesarean section
* Previous cesarean section
* Body mass index > 35 kg/m²

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Skin incision skewness | 10 minutes (from a photograph taken at the end of the operation)
  Skewness of the incision will be assessed using digital photos and an appropriate software.

SECONDARY OUTCOMES:
Incision length on both sides of the midline | 2 minutes (1 minute for measurement at the end of the operation and 1 minute postoperatively from a photo taken at the end of the operation)
  The length will be measured in cm.
Patient's perception of the scar | 1 minute (before discharge from hospital)
  Skewness and length of the scar are rated by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No